CLINICAL TRIAL: NCT05655351
Title: How Does Vaccination Against COVID-19 Affect Monocyte Production of Oxygenated Derivatives ?
Brief Title: Effect of a Vaccination Against COVID-19 on Monocyte Production of Oxygenated Derivatives.
Acronym: VACTICOV2
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NIMAO 2022-1; 2022-A02026-37 (Other: ANSM)
Record Dates: First submitted 2022-12-07; First posted 2022-12-19 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2024-09

CONDITIONS: CORONAVIRUS INFECTIONS
Keywords: COVID-19; Coronavirus; Anti-SARS-CoV-2 Vaccine; Reactive Oxygen Species
MeSH Terms: conditions — Coronavirus Infections; COVID-19 | interventions — Hematologic Tests

STUDY DESIGN:
Intervention Model Description: This is a pilot observational, single-center study with prospective longitudinal follow-up.
  Type of study: Non-Health Product. Category according to the Jarde law : Interventional research involving human subjects with minimal risks and constraints, Category 2.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients vaccinated with the anti-SARS-Cov-2 vaccination (Experimental): These patients will receive the anti-SARS-Cov-2 vaccination and their blood will be regularly monitored.
  Interventions: Biological: anti-SARS-Cov-2 vaccination

INTERVENTIONS:
Biological: anti-SARS-Cov-2 vaccination — For the purposes of the study, 10 mL of venous blood will be collected from each patient.
  Other Names: Blood test

SUMMARY:
Knowing that the vaccine antigen includes the ACE2 binding moiety (RBD), the hypothesis is that circulating vaccine antigen could reduce the enzymatic activity of ACE2, and thus increase circulating AngII concentration, monocyte ROS production and lymphocyte apoptosis. This hypothesis is supported by the fact that the Spike protein of SARSCoV-1, which uses the same receptor as SARS-CoV-2, induces a decrease in expression and activation of the Angiotensin II pathway in mice (Kuba et al. 2005).

DETAILED DESCRIPTION:
In this pandemic period, vaccination against SARSCoV- 2 is an essential weapon. However, the immune memory induced by current vaccines remains ephemeral, requiring early booster shots. It is primordial to improve this vaccine memory.

Recently it has been demonstrated that monocytes from certain individuals hospitalized for SARSCoV-2 infection spontaneously overproduced oxygenated derivatives (ROS) capable of inducing DNA damage in neighboring cells and T cell apoptosis (Kundura et al., 2022). In agreement with these observations, up to 50% of peripheral blood mononuclear cells (PBMC) from these patients showed DNA damage and its intensity was correlated with the percentage of apoptotic CD8+ T cells and lymphopenia.

Upon entry into the target cell, SARS-CoV-2 induces the internalization of its receptor, the protease Angiotensin Converting Enzyme 2 (ACE2), which is able to degrade Angiotensin II (AngII). Consequently, the circulating level of AngII was observed to be increased in some COVID-19 patients. It was also found that AngII induced monocyte ROS production via its receptor Angiotensin receptor 1 (AT1), making monocytes capable of damaging the DNA of co-cultured cells. Moreover, the plasma level of AngII in patients correlates with the level of ROS production and the ability to damage DNA of their monocytes. The level of anti SARS-CoV-2 antibodies was shown to be inversely correlated with the level of monocyte production of ROS production during the acute phase. This suggests that the activation cascade leading to lymphopenia described could damage the specific immune memory.

Now, a recent article has established the presence of circulating S1 vaccine antigen following the injection of an anti-SARS-CoV-2 vaccine with mRNA vaccine from D1 to D7 at a level of 68 ± 21 pg/mL (Ogata et al. 2022) similar to the level described in COVID-19 (Ogata et al. 2020). If the cascade of events we have identified is triggered by the circulation of the vaccine antigen, this could lead to could result in a reduced vaccine memory via lymphocyte apoptosis.

Knowing that the vaccine antigen includes the ACE2 binding moiety (RBD), the hypothesis is that circulating vaccine antigen could reduce the enzymatic activity of ACE2, and thus increase circulating AngII concentration, monocyte ROS production and lymphocyte apoptosis. This hypothesis is supported by the fact that the Spike protein of SARSCoV-1, which uses the same receptor as SARS-CoV-2, induces a decrease in expression and activation of the Angiotensin II pathway in mice (Kuba et al. 2005).

ELIGIBILITY:
Inclusion Criteria:

* Candidate for SARS-CoV-2 vaccination with an mRNA vaccine (Pfizer, Moderna).
* Subject has given free and informed consent.
* Subject who has signed the consent form.
* Person affiliated to or beneficiary of a health insurance plan.

Exclusion Criteria:

* Patients under treatment with N-acetylcysteine or sartan.
* Patients with a dysimmune pathology or immunosuppressive treatment.
* Person infected with SARS-CoV-2 within 3 months prior to inclusion.
* Person participating in a category 1 defined RIPH.
* Subject in an exclusion period as determined by another study.
* Person under court protection, guardianship or trusteeship.
* Subject who is unable to give consent.
* Subject for whom it is impossible to give clear information.
* Pregnant or breastfeeding woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-12-21 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Monocyte production of oxygenated derivatives (Reactive oxygen species) in patients under 30 years old before anti-SARS-CoV-2 vaccination with an mRNA vaccine. | Day 0
  The change (%) in the mean intensity of monocyte oxygen derivative (Reactive oxygen species) production will be measured by flow cytometry.
  All data will be collected on standardized electronic clinical report form available online.
  For ROS quantification: 106 PBMC will be re-suspended in 1μM dichloro-dihydro-fluorescein acetate (DCFH-DA) for 25minutes at room temperature. Data will be acquired on a Navios flow cytometer (Beckman Coulter) from 20,000 controlled events per sample and analyzed using Kaluza software (Kundura et al. 2022, in revision).
  The samples will be anonymized for blind measurement (at the Institute of Human Genetics in the team of Prof. Pierre Corbeau).
Monocyte production of oxygenated derivatives (Reactive oxygen species) in patients under 30 years old after anti-SARS-CoV-2 vaccination with an mRNA vaccine. | Day 7
  The change (%) in the mean intensity of monocyte oxygen derivative (Reactive oxygen species) production will be measured by flow cytometry.
  All data will be collected on standardized electronic clinical report form available online.
  For ROS quantification: 106 PBMC will be re-suspended in 1μM dichloro-dihydro-fluorescein acetate (DCFH-DA) for 25minutes at room temperature. Data will be acquired on a Navios flow cytometer (Beckman Coulter) from 20,000 controlled events per sample and analyzed using Kaluza software (Kundura et al. 2022, in revision).
  The samples will be anonymized for blind measurement (at the Institute of Human Genetics in the team of Prof. Pierre Corbeau).
Monocyte production of oxygenated derivatives (Reactive oxygen species) in patients under 30 years old after anti-SARS-CoV-2 vaccination with an mRNA vaccine. | Day 14
  The change (%) in the mean intensity of monocyte oxygen derivative (Reactive oxygen species) production will be measured by flow cytometry.
  All data will be collected on standardized electronic clinical report form available online.
  For ROS quantification: 106 PBMC will be re-suspended in 1μM dichloro-dihydro-fluorescein acetate (DCFH-DA) for 25minutes at room temperature. Data will be acquired on a Navios flow cytometer (Beckman Coulter) from 20,000 controlled events per sample and analyzed using Kaluza software (Kundura et al. 2022, in revision).
  The samples will be anonymized for blind measurement (at the Institute of Human Genetics in the team of Prof. Pierre Corbeau).
Monocyte production of oxygenated derivatives (Reactive oxygen species) in patients under 30 years old after anti-SARS-CoV-2 vaccination with an mRNA vaccine. | Day 28
  The change (%) in the mean intensity of monocyte oxygen derivative (Reactive oxygen species) production will be measured by flow cytometry.
  All data will be collected on standardized electronic clinical report form available online.
  For ROS quantification: 106 PBMC will be re-suspended in 1μM dichloro-dihydro-fluorescein acetate (DCFH-DA) for 25minutes at room temperature. Data will be acquired on a Navios flow cytometer (Beckman Coulter) from 20,000 controlled events per sample and analyzed using Kaluza software (Kundura et al. 2022, in revision).
  The samples will be anonymized for blind measurement (at the Institute of Human Genetics in the team of Prof. Pierre Corbeau).
Monocyte production of oxygenated derivatives (Reactive oxygen species) in patients aged 30 - 60 before anti-SARS-CoV-2 vaccination with an mRNA vaccine. | Day 0
  The change (%) in the mean intensity of monocyte oxygen derivative (Reactive oxygen species) production will be measured by flow cytometry.
  All data will be collected on standardized electronic clinical report form available online.
  For ROS quantification: 106 PBMC will be re-suspended in 1μM dichloro-dihydro-fluorescein acetate (DCFH-DA) for 25minutes at room temperature. Data will be acquired on a Navios flow cytometer (Beckman Coulter) from 20,000 controlled events per sample and analyzed using Kaluza software (Kundura et al. 2022, in revision).
  The samples will be anonymized for blind measurement (at the Institute of Human Genetics in the team of Prof. Pierre Corbeau).
Monocyte production of oxygenated derivatives (Reactive oxygen species) in patients aged 30 - 60 after anti-SARS-CoV-2 vaccination with an mRNA vaccine. | Day 7
  The change (%) in the mean intensity of monocyte oxygen derivative (Reactive oxygen species) production will be measured by flow cytometry.
  All data will be collected on standardized electronic clinical report form available online.
  For ROS quantification: 106 PBMC will be re-suspended in 1μM dichloro-dihydro-fluorescein acetate (DCFH-DA) for 25minutes at room temperature. Data will be acquired on a Navios flow cytometer (Beckman Coulter) from 20,000 controlled events per sample and analyzed using Kaluza software (Kundura et al. 2022, in revision).
  The samples will be anonymized for blind measurement (at the Institute of Human Genetics in the team of Prof. Pierre Corbeau).
Monocyte production of oxygenated derivatives (Reactive oxygen species) in patients aged 30 - 60 after anti-SARS-CoV-2 vaccination with an mRNA vaccine. | Day 14
  The change (%) in the mean intensity of monocyte oxygen derivative (Reactive oxygen species) production will be measured by flow cytometry.
  All data will be collected on standardized electronic clinical report form available online.
  For ROS quantification: 106 PBMC will be re-suspended in 1μM dichloro-dihydro-fluorescein acetate (DCFH-DA) for 25minutes at room temperature. Data will be acquired on a Navios flow cytometer (Beckman Coulter) from 20,000 controlled events per sample and analyzed using Kaluza software (Kundura et al. 2022, in revision).
  The samples will be anonymized for blind measurement (at the Institute of Human Genetics in the team of Prof. Pierre Corbeau).
Monocyte production of oxygenated derivatives (Reactive oxygen species) in patients aged 30 - 60 after anti-SARS-CoV-2 vaccination with an mRNA vaccine. | Day 28
  The change (%) in the mean intensity of monocyte oxygen derivative (ROS) production will be measured by flow cytometry.
  All data will be collected on standardized electronic clinical report form available online.
  For ROS quantification: 106 PBMC will be re-suspended in 1μM dichloro-dihydro-fluorescein acetate (DCFH-DA) for 25minutes at room temperature. Data will be acquired on a Navios flow cytometer (Beckman Coulter) from 20,000 controlled events per sample and analyzed using Kaluza software (Kundura et al. 2022, in revision).
  The samples will be anonymized for blind measurement (at the Institute of Human Genetics in the team of Prof. Pierre Corbeau).
Monocyte production of oxygenated derivatives (Reactive oxygen species) in patients aged over 60 before anti-SARS-CoV-2 vaccination with an mRNA vaccine. | Day 0
  The change (%) in the mean intensity of monocyte oxygen derivative (Reactive oxygen species) production will be measured by flow cytometry.
  All data will be collected on standardized electronic clinical report form available online.
  For ROS quantification: 106 PBMC will be re-suspended in 1μM dichloro-dihydro-fluorescein acetate (DCFH-DA) for 25minutes at room temperature. Data will be acquired on a Navios flow cytometer (Beckman Coulter) from 20,000 controlled events per sample and analyzed using Kaluza software (Kundura et al. 2022, in revision).
  The samples will be anonymized for blind measurement (at the Institute of Human Genetics in the team of Prof. Pierre Corbeau).
Monocyte production of oxygenated derivatives (Reactive oxygen species) in patients aged over 60 after anti-SARS-CoV-2 vaccination with an mRNA vaccine. | Day 7
  The change (%) in the mean intensity of monocyte oxygen derivative (Reactive oxygen species) production will be measured by flow cytometry.
  All data will be collected on standardized electronic clinical report form available online.
  For ROS quantification: 106 PBMC will be re-suspended in 1μM dichloro-dihydro-fluorescein acetate (DCFH-DA) for 25minutes at room temperature. Data will be acquired on a Navios flow cytometer (Beckman Coulter) from 20,000 controlled events per sample and analyzed using Kaluza software (Kundura et al. 2022, in revision).
  The samples will be anonymized for blind measurement (at the Institute of Human Genetics in the team of Prof. Pierre Corbeau).
Monocyte production of oxygenated derivatives (Reactive oxygen species) in patients aged over 60 after anti-SARS-CoV-2 vaccination with an mRNA vaccine. | Day 14
  The change (%) in the mean intensity of monocyte oxygen derivative (Reactive oxygen species) production will be measured by flow cytometry.
  All data will be collected on standardized electronic clinical report form available online.
  For ROS quantification: 106 PBMC will be re-suspended in 1μM dichloro-dihydro-fluorescein acetate (DCFH-DA) for 25minutes at room temperature. Data will be acquired on a Navios flow cytometer (Beckman Coulter) from 20,000 controlled events per sample and analyzed using Kaluza software (Kundura et al. 2022, in revision).
  The samples will be anonymized for blind measurement (at the Institute of Human Genetics in the team of Prof. Pierre Corbeau).
Monocyte production of oxygenated derivatives (Reactive oxygen species) in patients aged over 60 after anti-SARS-CoV-2 vaccination with an mRNA vaccine. | Day 28
  The change (%) in the mean intensity of monocyte oxygen derivative (Reactive oxygen species) production will be measured by flow cytometry.
  All data will be collected on standardized electronic clinical report form available online.
  For ROS quantification: 106 PBMC will be re-suspended in 1μM dichloro-dihydro-fluorescein acetate (DCFH-DA) for 25minutes at room temperature. Data will be acquired on a Navios flow cytometer (Beckman Coulter) from 20,000 controlled events per sample and analyzed using Kaluza software (Kundura et al. 2022, in revision).
  The samples will be anonymized for blind measurement (at the Institute of Human Genetics in the team of Prof. Pierre Corbeau).

SECONDARY OUTCOMES:
A) Plasma AngII level before anti-SARS-CoV-2 vaccination with an mRNA vaccine in patients aged under 30 | Day 0
  The AngII level before anti-SARS-CoV-2 vaccination with an mRNA vaccine will be measured by ELISA assay.
A) Plasma AngII level before anti-SARS-CoV-2 vaccination with an mRNA vaccine in patients aged 30 - 60 | Day 0
  The AngII level before anti-SARS-CoV-2 vaccination with an mRNA vaccine will be measured by ELISA assay.
A) Plasma AngII level before anti-SARS-CoV-2 vaccination with an mRNA vaccine in patients aged over 60 | Day 0
  The AngII level before anti-SARS-CoV-2 vaccination with an mRNA vaccine will be measured by ELISA assay.
A) Plasma AngII level after anti-SARS-CoV-2 vaccination with an mRNA vaccine in patients aged under 30 | Day 7
  The AngII level before anti-SARS-CoV-2 vaccination with an mRNA vaccine will be measured by ELISA assay.
A) Plasma AngII level after anti-SARS-CoV-2 vaccination with an mRNA vaccine in patients aged 30 - 60 | Day 7
  The AngII level before anti-SARS-CoV-2 vaccination with an mRNA vaccine will be measured by ELISA assay.
A) Plasma AngII level after anti-SARS-CoV-2 vaccination with an mRNA vaccine in patients aged over 60 | Day 7
  The AngII level before anti-SARS-CoV-2 vaccination with an mRNA vaccine will be measured by ELISA assay.
A) Plasma AngII level after anti-SARS-CoV-2 vaccination with an mRNA vaccine in patients aged under 30 | Day 14
  The AngII level before anti-SARS-CoV-2 vaccination with an mRNA vaccine will be measured by ELISA assay.
A) Plasma AngII level after anti-SARS-CoV-2 vaccination with an mRNA vaccine in patients aged 30 - 60 | Day 14
  The AngII level before anti-SARS-CoV-2 vaccination with an mRNA vaccine will be measured by ELISA assay.
A) Plasma AngII level after anti-SARS-CoV-2 vaccination with an mRNA vaccine in patients aged over 60 | Day 14
  The AngII level before anti-SARS-CoV-2 vaccination with an mRNA vaccine will be measured by ELISA assay.
A) Plasma AngII level after anti-SARS-CoV-2 vaccination with an mRNA vaccine in patients aged under 30 | Day 28
  The AngII level before anti-SARS-CoV-2 vaccination with an mRNA vaccine will be measured by ELISA assay.
A) Plasma AngII level after anti-SARS-CoV-2 vaccination with an mRNA vaccine in patients aged 30 - 60 | Day 28
  The AngII level before anti-SARS-CoV-2 vaccination with an mRNA vaccine will be measured by ELISA assay.
A) Plasma AngII level after anti-SARS-CoV-2 vaccination with an mRNA vaccine in patients aged over 60 | Day 28
  The AngII level before anti-SARS-CoV-2 vaccination with an mRNA vaccine will be measured by ELISA assay.
B) DNA lesion rate (%) and intensity in peripheral blood mononuclear cells (PBMC) before anti-SARS-CoV-2 mRNA vaccination in patients aged under 30 | Day 0
  Immunofluorescence measurement of the amount of γ-H2AX foci in PBMC as a percentage.
B) DNA lesion rate (%) and intensity in peripheral blood mononuclear cells (PBMC) before anti-SARS-CoV-2 mRNA vaccination in patients aged 30 - 60 | Day 0
  Immunofluorescence measurement of the amount of γ-H2AX foci in PBMC as a percentage.
B) DNA lesion rate (%) and intensity in peripheral blood mononuclear cells (PBMC) before anti-SARS-CoV-2 mRNA vaccination in patients aged over 60 | Day 0
  Immunofluorescence measurement of the amount of γ-H2AX foci in PBMC as a percentage.
B) DNA lesion rate (%) and intensity in peripheral blood mononuclear cells (PBMC) 7 days after anti-SARS-CoV-2 mRNA vaccination in patients aged under 30 | Day 7
  Immunofluorescence measurement of the amount of γ-H2AX foci in PBMC as a percentage.
B) DNA lesion rate (%) and intensity in peripheral blood mononuclear cells (PBMC) 7 days after anti-SARS-CoV-2 mRNA vaccination in patients aged 30 - 60 | Day 7
  Immunofluorescence measurement of the amount of γ-H2AX foci in PBMC as a percentage.
B) DNA lesion rate (%) and intensity in peripheral blood mononuclear cells (PBMC) 7 days after anti-SARS-CoV-2 mRNA vaccination in patients aged over 60 | Day 7
  Immunofluorescence measurement of the amount of γ-H2AX foci in PBMC as a percentage.
B) DNA lesion rate (%) and intensity in peripheral blood mononuclear cells (PBMC) 14 days after anti-SARS-CoV-2 mRNA vaccination in patients aged under 30 | Day 14
  Immunofluorescence measurement of the amount of γ-H2AX foci in PBMC as a percentage in patients aged under 30
B) DNA lesion rate (%) and intensity in peripheral blood mononuclear cells (PBMC) 14 days after anti-SARS-CoV-2 mRNA vaccination in patients aged 30 - 60 | Day 14
  Immunofluorescence measurement of the amount of γ-H2AX foci in PBMC as a percentage in patients aged under 30
B) DNA lesion rate (%) and intensity in peripheral blood mononuclear cells (PBMC) 14 days after anti-SARS-CoV-2 mRNA vaccination in patients aged over 60 | Day 14
  Immunofluorescence measurement of the amount of γ-H2AX foci in PBMC as a percentage in patients aged under 30
B) DNA lesion rate (%) and intensity in peripheral blood mononuclear cells (PBMC) 28 days after anti-SARS-CoV-2 mRNA vaccination in patients aged under 30 | Day 28
  Immunofluorescence measurement of the amount of γ-H2AX foci in PBMC as a percentage in patients aged under 30
B) DNA lesion rate (%) and intensity in peripheral blood mononuclear cells (PBMC) 28 days after anti-SARS-CoV-2 mRNA vaccination in patients aged 30 - 60 | Day 28
  Immunofluorescence measurement of the amount of γ-H2AX foci in PBMC as a percentage in patients aged under 30
B) DNA lesion rate (%) and intensity in peripheral blood mononuclear cells (PBMC) 28 days after anti-SARS-CoV-2 mRNA vaccination in patients aged over 60 | Day 28
  Immunofluorescence measurement of the amount of γ-H2AX foci in PBMC as a percentage in patients aged under 30
C) Rate of T cell apoptosis before anti-SARS-CoV-2 mRNA vaccination in patients aged under 30 | Day 0
  The percentage of T cells positive for annexin V (labelled with fluorescent annexin V) will be measured by flow cytometry
C) Rate of T cell apoptosis before anti-SARS-CoV-2 mRNA vaccination in patients aged 30 - 60 | Day 0
  The percentage of T cells positive for annexin V (labelled with fluorescent annexin V) will be measured by flow cytometry
C) Rate of T cell apoptosis before anti-SARS-CoV-2 mRNA vaccination in patients aged over 60 | Day 0
  The percentage of T cells positive for annexin V (labelled with fluorescent annexin V) will be measured by flow cytometry
C) Rate of T cell apoptosis 7 days after anti-SARS-CoV-2 mRNA vaccination in patients aged under 30 | Day 7
  The percentage of T cells positive for annexin V (labelled with fluorescent annexin V) will be measured by flow cytometry
C) Rate of T cell apoptosis 7 days after anti-SARS-CoV-2 mRNA vaccination in patients aged 30 - 60 | Day 7
  The percentage of T cells positive for annexin V (labelled with fluorescent annexin V) will be measured by flow cytometry
C) Rate of T cell apoptosis 7 days after anti-SARS-CoV-2 mRNA vaccination in patients aged over 60 | Day 7
  The percentage of T cells positive for annexin V (labelled with fluorescent annexin V) will be measured by flow cytometry
C) Rate of T cell apoptosis 14 days after anti-SARS-CoV-2 mRNA vaccination in patients aged under 30 | Day 14
  The percentage of T cells positive for annexin V (labelled with fluorescent annexin V) will be measured by flow cytometry
C) Rate of T cell apoptosis 14 days after anti-SARS-CoV-2 mRNA vaccination in patients aged 30 - 60 | Day 14
  The percentage of T cells positive for annexin V (labelled with fluorescent annexin V) will be measured by flow cytometry
C) Rate of T cell apoptosis 14 days after anti-SARS-CoV-2 mRNA vaccination in patients aged over 60 | Day 14
  The percentage of T cells positive for annexin V (labelled with fluorescent annexin V) will be measured by flow cytometry
C) Rate of T cell apoptosis 28 days after anti-SARS-CoV-2 mRNA vaccination in patients aged under 30 | Day 28
  The percentage of T cells positive for annexin V (labelled with fluorescent annexin V) will be measured by flow cytometry
C) Rate of T cell apoptosis 28 days after anti-SARS-CoV-2 mRNA vaccination in patients aged 30 - 60 | Day 28
  The percentage of T cells positive for annexin V (labelled with fluorescent annexin V) will be measured by flow cytometry
C) Rate of T cell apoptosis 28 days after anti-SARS-CoV-2 mRNA vaccination in patients aged over 60 | Day 28
  The percentage of T cells positive for annexin V (labelled with fluorescent annexin V) will be measured by flow cytometry
D) Presence of lymphopenia before anti-SARS-CoV-2 vaccination by an mRNA vaccine in patients aged under 30 | Day 0
  Complete blood count. Lymphocytes will be measured as a percentage.
D) Presence of lymphopenia before anti-SARS-CoV-2 vaccination by an mRNA vaccine in patients aged 30 - 60 | Day 0
  Complete blood count. Lymphocytes will be measured as a percentage.
D) Presence of lymphopenia before anti-SARS-CoV-2 vaccination by an mRNA vaccine in patients aged over 60 | Day 0
  Complete blood count. Lymphocytes will be measured as a percentage.
D) Presence of lymphopenia 7 days after anti-SARS-CoV-2 vaccination by an mRNA vaccine in patients aged under 30 | Day 7
  Complete blood count. Lymphocytes will be measured as a percentage.
D) Presence of lymphopenia 7 days after anti-SARS-CoV-2 vaccination by an mRNA vaccine in patients aged 30 - 60 | Day 7
  Complete blood count. Lymphocytes will be measured as a percentage.
D) Presence of lymphopenia 7 days after anti-SARS-CoV-2 vaccination by an mRNA vaccine in patients aged over 60 | Day 7
  Complete blood count. Lymphocytes will be measured as a percentage.
D) Presence of lymphopenia 14 days after anti-SARS-CoV-2 vaccination by an mRNA vaccine in patients aged under 30 | Day 14
  Complete blood count. Lymphocytes will be measured as a percentage.
D) Presence of lymphopenia 14 days after anti-SARS-CoV-2 vaccination by an mRNA vaccine in patients aged 30 - 60 | Day 14
  Complete blood count. Lymphocytes will be measured as a percentage.
D) Presence of lymphopenia 14 days after anti-SARS-CoV-2 vaccination by an mRNA vaccine in patients aged over 60 | Day 14
  Complete blood count. Lymphocytes will be measured as a percentage.
D) Presence of lymphopenia 28 days after anti-SARS-CoV-2 vaccination by an mRNA vaccine in patients aged under 30 | Day 28
  Complete blood count. Lymphocytes will be measured as a percentage.
D) Presence of lymphopenia 28 days after anti-SARS-CoV-2 vaccination by an mRNA vaccine in patients aged 30 - 60 | Day 28
  Complete blood count. Lymphocytes will be measured as a percentage.
D) Presence of lymphopenia 28 days after anti-SARS-CoV-2 vaccination by an mRNA vaccine in patients aged over 60 | Day 28
  Complete blood count. Lymphocytes will be measured as a percentage.
E) Quantification of anti-S antibodies in patients aged under 30 before anti-SARS-CoV-2 vaccination with an mRNA vaccine. | Day 0
  Anti-S antibodies will be quantified by enzyme-linked immunosorbent assay (ELISA) in Antibody Units/mL
E) Quantification of anti-S antibodies in patients aged 30 - 60 before anti-SARS-CoV-2 vaccination with an mRNA vaccine. | Day 28
  Anti-S antibodies will be quantified by enzyme-linked immunosorbent assay (ELISA) in Antibody Units/mL
E) Quantification of anti-S antibodies in patients aged over 60 before anti-SARS-CoV-2 vaccination with an mRNA vaccine. | Day 28
  Anti-S antibodies will be quantified by enzyme-linked immunosorbent assay (ELISA) in Antibody Units/mL
F) Constitution of a biobank | Day 28
  Plasma and cell samples will be referenced and stored for use in future studies.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nîmes, Hôpital Universitaire Caremeau, Nîmes, France, France

REFERENCES:
- [Result] Gimenez S, Hamrouni E, Andre S, Picard M, Soundaramourty C, Lozano C, Vincent T, Tran TA, Kundura L, Estaquier J, Corbeau P. Monocytic reactive oxygen species-induced T-cell apoptosis impairs cellular immune response to SARS-CoV-2 mRNA vaccine. J Allergy Clin Immunol. 2025 May;155(5):1635-1646. doi: 10.1016/j.jaci.2025.01.003. Epub 2025 Jan 10. PMID 39800264